CLINICAL TRIAL: NCT03278015
Title: Phase 2 Trial of Gemcitabine vs S-1 vs Gemcitabine Plus Nab-paclitaxel as Adjuvant Chemotherapy of Post-operative Pancreatic Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dabin Xu, Associate Chief Doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XDB-001
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Cancer of Pancreas
Keywords: S-1; nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nab-paclitaxel plus Gemcitabine (Experimental): Nanoparticle albumin-bound paclitaxel is given at 100mg/m2 intravenously over 30 minutes in combination with Gemcitabine 1000mg/m2 intravenously on day 1 and 8 of each 21-days cycle. Number of cycle: 6 cycles.
  Interventions: Drug: Nab-paclitaxel plus Gemcitabine
- Gemcitabine monotherapy (Experimental): Gemcitabine is given at 1000mg/m2 intravenously on day 1 and 8 of each 21-days cycle. Number of cycle: 6 cycles.
  Interventions: Drug: Gemcitabine monotherapy
- S-1 monotherapy (Experimental): S-1 is orally administered (40-60 mg according to the body surface, Bid) on day 1-14 of each 21-days cycle. Number of cycle: 6 cycles.
  Interventions: Drug: S-1 monotherapy

INTERVENTIONS:
Drug: Nab-paclitaxel plus Gemcitabine — Nanoparticle albumin-bound paclitaxel is given at 100mg/m2 intravenously over 30 minutes in combination with Gemcitabine 1000mg/m2 intravenously on day 1 and 8 of each 21-days cycle. Number of cycle: 6 cycles.
  Other Names: nab-paclitaxel abraxane ABI-007; GEMXAR
  Arms: Nab-paclitaxel plus Gemcitabine
Drug: Gemcitabine monotherapy — Gemcitabine is given at 1000mg/m2 intravenously on day 1 and 8 of each 21-days cycle. Number of cycle: 6 cycles.
  Other Names: GEMXAR
  Arms: Gemcitabine monotherapy
Drug: S-1 monotherapy — S-1 is orally administered (40-60 mg according to the body surface, Bid) on day 1-14 of each 21-days cycle. Number of cycle: 6 cycles.
  Arms: S-1 monotherapy

SUMMARY:
Pancreatic cancer is one of the deadliest tumor types, there is no effective treatment method clinically. Recently radical surgical resection is recommended for this cancer, How to improve the survival rate of patients is the doctors' goals . Postoperative chemotherapy can partly raise post-operative survival rate. the purpose of this study is to three chemotherapy regimens(gemcitabine monotherapy, S-1 monotherapy and combining nab-paclitaxel with gemcitabine),which is best regimens for raising patients' survival rate, and will provide a chemotherapy choice for clinic therapy of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form.
2. Man or woman aged 18 years to 80 years.
3. Histologically confirmed pancreatic carcinoma, and the histological type is ductal adenocarcinoma.
4. Mild (Child-Pugh A), moderate (Child-Pugh B) and some preferable severe (Child-Pugh C, <=10) hepatic dysfunction according to the Child-Pugh Scoring system criteria.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-3, with life expectation of no less than 12 weeks.
6. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥1.5 x 109/L; platelets ≥ 70 x 109/L; hemoglobin ≥ 8.0 g/dL.
7. Albumin ≥ 30 g/L.
8. Adequate hepatic function as evidenced by Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN); Serum total bilirubin ≤ 1.5 x ULN; Serum creatinine ≤ 1.5 x ULN.
9. Females of childbearing potential must have a negative serum pregnancy test and must not breast-feed before the first dose. Male also need contraception.
10. Willing and able to comply with study procedures for the duration of the study.

Exclusion Criteria:

1. Hypertension, and unable to drop to normal level (systolic pressure >140 mmHg, diastolic pressure >90 mmHg) after treatment.
2. Patients have active cardiac disease including any of the following:

   1. In resting state, average correction QTc > 470 msec on mean value of 3 times screening ECGs.
   2. Any clinically significant abnormal ECG form, for example, complete left bundle branch block, 3-degree atrioventricular block, 2-degree atrioventricular block, or PR interval > 250 msec.
   3. Any factors may increase the risk of QTc prolongation or arrhythmic event.
   4. Left ventricular ejection fraction (LVEF) < 50%.
3. Patient weight still in losing period.
4. History of gastrointestinal bleeding or a gastrointestinal bleeding tendency, such as esophageal varices with high risk of bleeding, local active ulcerative lesions, fecal occult blood test>= (+ +) within the past 6 months, shall not enter the trial. If fecal occult blood test (+), the patient is requested for gastroscopy.
5. Patients with abdominal fistula, gastrointestinal perforation or abdominal abscess within the past 28 days, should not enter the trial.
6. Patients with coagulant function abnormality (INR > 1.5 or prothrombin time (PT) > ULN + 4 sec), with bleeding tendency or are treated with thrombolytic or anticoagulant therapy.
7. Patients with unstable or serious concurrent medical conditions are excluded. The researcher evaluates that the patient who is not suitable for participation in the study. Patients with active infection, for example, HBV, HCV, or HIV.
8. Uncontrollable nausea, vomit, chronic gastrointestinal disorders leading to unable to swallow drugs, which may affect the fully absorption of S-1.
9. Patients with mental illness, or with psychiatric history of drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival(DFS) | 3 years
  To determine the DFS of post-operative patients with pancreatic cancer
overall survival time (OS) | 5 years
  To determine the OS post-operative patients with pancreatic cancer
median overall survival time (mOS) | 5 years
  To determine the mOS post-operative patients with pancreatic cancer

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 3 years
  All patients must be considered in response analysis, including those who discontinue treatment or who die for any reason prior to response evaluations
Quality of Life Assessment | 3 years
safety profile | 3 years
  Treatment-emergent adverse events, drug-related adverse events will be analysed by 3 groups
Disease control rate(DCR) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China